CLINICAL TRIAL: NCT04681430
Title: Reconvalescent Plasma / Camostat Mesylate Early in Sars-CoV-2 Q-PCR (COVID-19) Positive High-risk Individuals
Brief Title: Reconvalescent Plasma/Camostat Mesylate Early in SARS-CoV-2 Q-PCR (COVID-19) Positive High-risk Individuals
Acronym: RES-Q-HR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: The Federal Ministry of Health, Germany (Bundesministerium für Gesundheit, BMG) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RES-Q-HR; 2020-004695-18 (EudraCT Number)
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Corona Virus Infection; SARS-CoV-2 Infection; SARS-CoV-2 PCR Test Positive; SARS-CoV-2 Acute Respiratory Disease
Keywords: SARS-CoV-2; Covid-19; camostat mesilate; reconvalescent plasma; TMPRSS2
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — camostat; Standard of Care

STUDY DESIGN:
Intervention Model Description: The study is a multicenter trial that will be conducted in approx. 10 - 15 centers in Germany.
  At each center, patients will be randomized into four groups: two treatment groups and two control groups. The randomization rate in this study is two to one (2:1) in favor to therapy, i.e.
  included patients have twice the chance to receive interventional therapy than placebo / SoC.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The camostat mesylate and its placebo group will be double blinded while the CP and its placebo will be open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- convalescent plasma (CP) (Experimental): Administration of 2 units of CP (neutralizing anti-SARS-CoV-2 antibody titer of at least 1:160) on day 1
  Interventions: Biological: Convalescent plasma
- Standard of Care (Other): Standard of care allowed
  Interventions: Other: Standard of Care (SoC)
- Camostat Mesilate (Experimental): Tablets 600 mg per day in 3 doses over 7 days
  Interventions: Drug: Camostat Mesilate
- Placebo camostat (Placebo Comparator): Placebo Tablets in 3 doses over 7 days (blinded)
  Interventions: Drug: Placebo for Camostat Mesilate

INTERVENTIONS:
Biological: Convalescent plasma — transfusion of convalescent plasma (CP) with neutralizing antibodies against anti-SARS-CoV-2 ((titer of at least 1:160)
  Arms: convalescent plasma (CP)
Drug: Camostat Mesilate — Tablets over 7 days, daily dose of 600 mg split into 3 doses
  Arms: Camostat Mesilate
Drug: Placebo for Camostat Mesilate — Placebo Tablets over 7 days, split into 3 doses
  Arms: Placebo camostat
Other: Standard of Care (SoC) — Control Arm for convalescent plasma (CP)
  Arms: Standard of Care

SUMMARY:
This study is a 4-arm, multicenter, randomized, partly double- blind, controlled trial to evaluate the safety and efficacy of convalescent serum (CP) or camostat mesylate with control or placebo in adult patients diagnosed with SARS-CoV-2 and high risk for moderate/severe COVID-19. The working hypothesis to be tested in the RES-Q-HR study is that the early use of convalescent plasma (CP) or camostat mesylate (Foipan®) reduces the likelihood of disease progression to modified WHO stages 4b-8 in SARS-CoV-2 positive adult patients at high risk of moderate or severe COVID-19 progression. The primary endpoint of the study is the cumulative number of individuals who progressed to or beyond category 4b on the modified WHO (World Health Organization) COVID-19 ordinal scale within 28 days after randomization.

DETAILED DESCRIPTION:
The novel coronavirus designated SARS CoV-2, and the disease caused by this virus designated COVID-19. No treatment is available for early disease stages and non-hospitalized patients to date. This trial focusses on SARS-CoV-2 positive patients with pre-existing risk factors for a moderate or severe COVID-19 disease course. This study is a 4-arm, multicenter, randomized, partly double-blind, controlled trial to evaluate the safety and efficacy of convalescent serum (CP) or camostat mesylate with control or placebo in adult patients diagnosed with SARS-CoV-2 and high risk for moderate/severe COVID-19. Camostat mesylate acts as an inhibitor of the host cell serine protease TMPRSS2 and prevents the virus from entering the cell. Convalescent plasma (CP) represents another antiviral strategy in terms of passive immunization. The working hypothesis to be tested in the RES-Q HR study is that the early use of convalescent plasma (CP) or camostat mesylate (Foipan®) reduces the likelihood of disease progression to modified WHO stages 4b-8 in SARS-CoV-2 positive adult patients at high risk of moderate or severe COVID-19 progression.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals (female, male, diverse) ≥ 18 years with SARS-CoV-2 infection, confirmed by PCR before study enrollment
2. SARS-CoV-2 positive PCR ≤ 3 days old (date of NP swab)
3. Presence of ≥ 1 SARS-CoV-2 typical symptom (fever, cough, shortness of breath, sore throat, headache, fatigue, smell/and or taste disorder, diarrhea, abdominal symptoms, exanthema) and symptom duration <= 3 days.
4. Ability to provide written informed consent
5. Presence of at least one of the following criteria:

   * Patients > 75 years
   * Patients > 65 years with at least one other risk factor (BMI >35 kg/m2, coronary artery disease, chronic kidney disease (CKD) with glomerular filtration rate (GFR) <60 ml/min but >= 30 ml/min, diabetes mellitus, active tumor disease)
   * Patients with a BMI >35 kg/m2 with at least one other risk factor (CAD, CKD with GFR <60 ml/min but >= 30 ml/min, diabetes mellitus, active tumor disease)
   * Patients with a BMI >40 kg/m2
   * Patients with chronic obstructive pulmonary disease (COPD) and/or pulmonary fibrosis

Exclusion Criteria:

1. Age <18 years
2. Unable to give informed consent
3. Pregnant women or breast-feeding mothers
4. Previous transfusion reaction or other contraindication to a plasma transfusion
5. Known hypersensitivity to camostat mesylate and/or severe pancreatitis
6. Volume stress due to CP administration would be intolerable
7. Known IgA deficiency
8. Life expectancy < 6 months
9. Duration SARS-CoV-2 typical symptoms > 3 days
10. SARS-CoV-2 PCR detection older than 3 days
11. SARS-CoV-2 associated clinical condition >= WHO stage 3 (patients hospitalized for other reasons than COVID-19 may be included if they fulfill all inclusion and none of the exclusion criteria).
12. Previously or currently hospitalized due to SARS-CoV-2
13. Previous antiviral therapy for SARS-CoV-2
14. alanine aminotransferase (ALT) or aspartate transferase (AST) > 5 times upper limit of normal (ULN) at screening
15. Liver cirrhosis > Child A (patients with Child B/C cirrhosis are excluded from the trial)
16. Chronic kidney disease with GFR < 30 ml/min
17. Concurrent or planned anticancer treatment during trial period
18. Accommodation in an institution due to legal orders (§40(4) AMG).
19. Any psycho-social condition hampering compliance with the study protocol.
20. Evidence of current drug or alcohol abuse.
21. Use of other investigational treatment within 5 half-lives of enrollment is prohibited
22. Previous use of convalescent plasma for COVID-19
23. Concomitant proven influenza A infection
24. Patients with organ or bone marrow transplant in the three months prior to Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
WHO ordinal Covid-19 scale up to day 28 | up to and including day 28
  The primary endpoint of the study is the number of individuals whose clinical status is on the COVID-19 modified WHO ordinal scale ≥ 4b up to and including day 28

SECONDARY OUTCOMES:
Cumulative number WHO categories 4b-8 | day 8, day 14, day 56 and day 90
  Cumulative number of persons in the respective treatment arms versus SoC/placebo in WHO categories 4b-8
Cumulative number WHO categories 3-4a | day 8, day 14, day 28, day 56 and day 90
  Cumulative number of persons in the respective treatment arms versus SoC/placebo in WHO categories 3-4a
Not hospitalized | at day 90
  Cumulative number of participants not hospitalized at day 90
All-cause mortality | at day 90
  All-cause mortality at day 90
Reinfection | up to day 90
  Number of patient with SARS-CoV-2 reinfection up to day 90
Secondary sclerosing cholangitis (SSC) | at day 90
  Number of patient with secondary sclerosis cholangitis at day 90
chronic pulmonary disease as sequelae from COVID-19 | at day 90
  Number of patient with COVID-19 associated chronic pulmonary disease
patients with remdesivir treatment | up to day 90
  The proportion of patients with remdesivir therapy
COVID-19 WHO status of patients at start of remdesivir treatment | up to day 90
  The clinical status on the WHO COVID-19 ordinal scale of at the start of remdesivir treatment WHO ordinal scale ranges from 0 to 8; whereas 0 = no COVID-19 infection and 8 = death
patients with dexamethasone treatment | up to day 90
  The proportion of patients on dexamethasone therapy
COVID-19 WHO status of patients at start of dexamethasone treatment | up to day 90
  The clinical status on the WHO COVID-19 ordinal scale of at the start of dexamethasone treatment
  WHO ordinal scale ranges from 0 to 8; whereas 0 = no COVID-19 infection and 8 = death
resolution of COVID-19 symptoms | until day of resolution up to day 90
  Time to resolution of COVID-19 related symptoms (e.g. fever)
negative SARS-CoV-2-PCR test | until day of first negative test up to day 90
  Time to first negative SARS-CoV-2-PCR (polymerase chain reaction)
Oxygen therapy | number of days with oxygen therapy up to day 90
  Duration of oxygen therapy (in days)
COVID-19 pneumonia | up to day 90
  Frequency of occurrence of COVID-19 pneumonia
Percentage of participants requiring mechanical ventilation | up to day 90
  Percentage of participants in each group with need for mechanical ventilation
Number of ventilation days per participant up to day 90 | up to day 90
  Number of ventilation days per participant up to day 90
hospital stay and intensive care | up to day 90
  Duration of hospital stay (in days), duration in intensive care/intermediate care (IMC) (in days)
Mortality | at day 28
  All-cause mortality at day 28
SAEs | up to day 90
  Cumulative incidence of Serious Adverse Events (SAE) per group within 90 days follow up
Grade 3/4 AEs | up to day 90
  Cumulative incidence of grade 3/4 Adverse Events (AE) per group
SARS-CoV-2 antibody IgA concentrations | on day 8, day 14, day 90
  SARS-CoV-2 antibody concentrations (IgA in g/l) in serum on day 8, day 14, day 90
SARS-CoV-2 antibody IgG concentrations | on day 8, day 14, day 90
  SARS-CoV-2 antibody concentrations (IgG in g/l) in serum on day 8, day 14, day 90
SARS-CoV-2 neutralizing antibody titers | on day 8, day 14, day 90
  SARS-CoV-2 neutralizing antibody titers in serum on day 8, day 14, day 90
Plasma treatment screening failures | up to day 8 (End of treatment)
  Number of screening failures due to the lack of a suitable plasma preparation

CONTACTS AND LOCATIONS:
Overall Officials: Verena Keitel-Anselmino, Prof.Dr.med., Principal Investigator — Klinik für Gastroenterologie, Hepatologie und Infektiologie Universitätsklinikum Düsseldorf
Locations (6):
- Germany (6):
  - Abteilung Infektiologie Klinik für Innere Medizin II Department Innere Medizin Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinik und Poliklinik für Innere Medizin II Klinikum rechts der Isar Technische Universität München, München, Bavaria
  - Universitätsklinikum Frankfurt Medizinische Klinik 2: Hämatologie, Onkologie, Hämostaseologie, Rheumatologie, Infektiologie/HIV, Frankfurt am Main, Hesse
  - Klinikum Dortmund, Dortmund, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf Klinik für Hepatologie und Infektiologie, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keitel V, Jensen B, Feldt T, Fischer JC, Bode JG, Matuschek C, Bolke E, Budach W, Plettenberg C, Scheckenbach K, Kindgen-Milles D, Timm J, Muller L, Kolbe H, Stohr A, Calles C, Hippe A, Verde P, Spinner CD, Schneider J, Wolf T, Kern WV, Nattermann J, Zoufaly A, Ohmann C, Luedde T; RES-Q-HR Trial Team. Reconvalescent plasma/camostat mesylate in early SARS-CoV-2 Q-PCR positive high-risk individuals (RES-Q-HR): a structured summary of a study protocol for a randomized controlled trial. Trials. 2021 May 17;22(1):343. doi: 10.1186/s13063-021-05181-0. PMID 34001215